CLINICAL TRIAL: NCT00060398
Title: Study Of Epoetin Alfa Vs Epoetin Alfa With Dexamethasone In Hormone Refractory Prostate Cancer Patients: Impact On Fatigue, Anemia, Functional Status And Quality Of Life
Brief Title: Epoetin Alfa With or Without Dexamethasone in Treating Fatigue and Anemia in Patients With Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000301881; ECOG-E1Z01
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Anemia; Fatigue; Prostate Cancer
Keywords: recurrent prostate cancer; anemia; fatigue
MeSH Terms: conditions — Anemia; Fatigue; Prostatic Neoplasms | interventions — Epoetin Alfa; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: epoetin alfa
Drug: dexamethasone

SUMMARY:
RATIONALE: Epoetin alfa may stimulate red blood cell production and may help improve cancer-related anemia and fatigue. Steroid therapy with dexamethasone may increase the effectiveness of epoetin alfa. It is not yet known if epoetin alfa is more effective with or without dexamethasone in treating anemia-related fatigue in patients with prostate cancer.

PURPOSE: This randomized phase III trial is studying epoetin alfa and dexamethasone to see how well they work compared to epoetin alfa alone in treating anemia-related fatigue in patients with prostate cancer that is refractory to treatment with hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of epoetin alfa with or without dexamethasone on the level of cancer-related fatigue measured by the FACIT fatigue subscale, in patients with hormone-refractory prostate cancer.
* Compare the effect of these regimens on increasing hemoglobin levels in these patients.
* Compare the effect of these regimens on palliation of other disease-related symptoms and on functional status and overall quality of life of these patients.
* Compare the survival rate of these regimens in these patients.
* Compare the toxicity profile of these regimens in these patients.
* Determine the incidence of adrenal suppression in these patients after receiving dexamethasone therapy.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to usual fatigue severity on the Brief Fatigue Inventory numerical scale (3-6 vs 7-10) and hemoglobin level (8-10 g/dL vs 10.1-11.9 g/dL). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive epoetin alfa subcutaneously once a week.
* Arm II: Patients receive epoetin alfa as in arm I and oral dexamethasone once a day.

In both arms, treatment continues for 12 weeks in the absence of unacceptable toxicity.

Quality of life and fatigue are assessed at baseline and then at 4, 8, and 12 weeks.

Patients are followed for 3 years.

PROJECTED ACCRUAL: A total of 282 patients (141 per treatment arm) will be accrued for this study within approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * Hormone-refractory disease as evidenced by progression on bone scan or CT scan with a rising prostate-specific antigen
* Prior bilateral orchiectomy OR other primary hormonal therapy (e.g., estrogen therapy or luteinizing hormone-releasing hormone analog [LHRH] and flutamide) with evidence of treatment failure

  * Concurrent continual LHRH agonist therapy (e.g., depot leuprolide or goserelin) required for patients who have not undergone bilateral orchiectomy
* Must have anemia with hemoglobin ≥ 8 g/dL and < 12 g/dL within the past 14 days
* Must be iron replete (i.e., ferritin > 50 ng/mL) within the past 30 days
* Presence of fatigue with usual fatigue severity ≥ 3 on the 0-10 numerical scale of the Brief Fatigue Inventory within the past 14 days

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-3

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics
* No disseminated intravascular coagulation
* No autoimmune hemolytic anemia

Hepatic

* AST and ALT ≤ 2 times upper limit of normal
* No prior hemochromatosis or iron intolerance

Renal

* Creatinine < 2.5 mg/dL

Cardiovascular

* Adequate blood pressure (i.e., systolic blood pressure < 140 mm Hg and diastolic blood pressure < 90 mm Hg) (treated or untreated)
* No history of thromboembolic events
* No unstable angina
* No poorly controlled cardiac disease

Other

* Fertile patients must use effective contraception
* Able to read, understand, and answer questions on the symptom and quality of life study instruments
* No ongoing chronic hemorrhage (e.g., gross hematuria due to advanced prostate cancer)* NOTE: *Microscopic hematuria allowed
* No acute or subacute illness that may require transfusion
* No gastrointestinal bleeding
* No active systemic infection
* No known or suspected hypersensitivity to human albumin
* No known or suspected hypersensitivity to mammalian cell-derived products
* No uncontrolled diabetes

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 30 days since prior epoetin alfa

Chemotherapy

* More than 21 days since prior chemotherapy
* No more than 2 different types of prior chemotherapy regimens for hormone-refractory prostate cancer

Endocrine therapy

* See Disease Characteristics
* More than 30 days since prior corticosteroids for hormone-refractory prostate cancer

  * Episodic use of low-dose steroids for other causes is allowed

Radiotherapy

* More than 21 days since prior radiotherapy
* Concurrent radiotherapy allowed

Surgery

* See Disease Characteristics

Other

* More than 8 weeks since prior blood transfusion
* No concurrent oral or intravenous antibiotics

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2004-09-29 (Actual); Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Fatigue response as measured by the Functional Assessment of Chronic Illness Therapy Fatigue Subscale

SECONDARY OUTCOMES:
Anemia response at 3 months
Functional level as measured by the Functional Assessment of Cancer Therapy-General Scale and Brief Fatigue Inventory functional interference score monthly
Symptom distress as measured by the Memorial Symptom Assessment Scale-Short Form and the number of symptoms monthly
Quality of life as measured by the Functional Assessment of Cancer Therapy-General Scale monthly
Survival at 6 months
Adrenal suppression
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Shirley S. Hwang, RN, MS, Study Chair — Veterans Affairs Medical Center - East Orange
Locations (140):
- United States (140):
  - Memorial Medical Center Cancer Services, Modesto, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Northwest Medical Specialist, PC, Niles, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Midwest Cancer Research Group, Incorporated, Skokie, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - McFarland Clinic, P. C., Ames, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, P.A. - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, P.A. - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, P.A. - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, P.A. - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, P.A. - Salina, Salina, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Lawrence Memorial Hospital of Medford, Medford, Massachusetts
  - Commonwealth Hematology-Oncology P. C. - Quincy, Quincy, Massachusetts
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - Shore Memorial Hospital - Somers Point, Somers Point, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Dean Medical Center - Fish Hatchery, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin